CLINICAL TRIAL: NCT02157259
Title: An Observational Study of the Causes, Management, and Outcomes of Community-acquired Sepsis and Severe Sepsis in Southeast Asia
Acronym: SEA050
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); FHI 360 (Other); Social & Scientific Systems Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SEA-050 Sepsis Study
Record Dates: First submitted 2014-05-20; First posted 2014-06-05 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Sepsis; Severe Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study to identify the etiology, management, and outcome of community-acquired sepsis and severe sepsis in children and adults in Southeast Asia. The study will take place in Thailand, Vietnam, and Indonesia, the partner countries of SEAICRN. Potential study patients will be any patients (both children and adults) who are presented at the hospital with community-acquired sepsis or severe sepsis and require hospitalization.

DETAILED DESCRIPTION:
The study will enroll 2,250 total patients with sepsis or severe sepsis patients up to 2 years of study. 750 patients will be enrolled in each of Thailand, Vietnam, and Indonesia. There will be 3 sites in each country and some sites will function as cluster/unit sites linking up to 3 hospitals as one 'site' to enable adequate enrollment of both adult and pediatric cases.

Primary objective of the study is to determine the causes of community-acquired sepsis and severe sepsis in adult and pediatric subjects across Southeast Asia.

The secondary objectives are as follow:

* To define the current acute management (within the first 48 hours after admission) of subjects presenting with community-acquired sepsis and severe sepsis and gaps of current practice as defined by the surviving sepsis campaign 2012. This will provide the basis for designing practical interventions to reduce the mortality of subjects with sepsis and severe sepsis in the future.
* To define the clinical outcomes of community-acquired sepsis and severe sepsis in Southeast Asia.
* To identify risk factors associated with sepsis or severe sepsis.
* To determine the extent of antimicrobial resistance in organisms that cause community-acquired sepsis and severe sepsis in Southeast Asia and to determine the association between antimicrobial resistance and mortality.
* To evaluate the accuracy of selected rapid diagnostic tests (RDTs) in determining the causes of community-acquired sepsis and severe sepsis compared to well-defined gold standard tests.

As this is an observational study and not a clinical trial, researchers will not be involved in the management, care and treatment of study subjects. This will remain the responsibility of the attending medical staff according to standard of care (SOC) in the participating hospitals. Therefore the research study will not influence patient management. SOC for sepsis and severe sepsis in each subject will be recorded, and will be reported as summary statistics at the end of the study. This will not be used to influence the management and care of sepsis and severe sepsis cases at the participating hospitals during the study period, but will be used to guide the improvement of the SOC after the study is complete.

NOTE: EACH INSTITUTION IN THIS STUDY IS ITS OWN SPONSOR AS LISTED BELOW:

1. Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand.
2. Queen Sirikit National Institute of Child Health, Bangkok, Thailand.
3. Children's Hospital 1 Ho Chi Minh City, Vietnam.
4. Children's Hospital 2 Ho Chi Minh City, Vietnam.
5. Hospital for Tropical Diseases Ho Chi Minh City, Vietnam.
6. National Hospital for Pediatrics Hanoi, Vietnam.
7. National Hospital for Tropical Diseases, Hanoi, Vietnam.
8. Hue Central Hospital, Hue City, Vietnam.
9. Dr. Wahidin Soedirohusodo Hospital Makassar, Indonesia.
10. Dr. Sardjito Hospital Yogyakarta, Indonesia.
11. Dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia
12. Sappasithiprasong Hospital Ubonratchathani, Thailand
13. Chiangrai Prachanukroh Hospital, Chiangrai Thailand
14. University of Oxford, United Kingdom

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥30 days old and weighing at least 3 kg or more on the day of enrollment into the study
2. Required hospitalization as decided by the attending physician
3. Documented by attending physician that an infection is the primary cause of illness leading to the hospitalization. These can be infections due to any pathogens (bacteria, viruses, fungi and parasites).
4. Presence of Systemic Inflammatory Response Syndrome (SIRS):

   4.1 For adults (≥ 18 years old), any combination of a minimum of any 3 of the following 20 parameters
   * Fever or hypothermia (Core body temperature defined as >38.3 C or <36.0 C)
   * Tachycardia (heart rate >90 beats per minute)
   * Tachypnea (respiratory rate >20 per minute)
   * Arterial hypotension (systolic blood pressure (SBP) <90 mmHg, mean arterial pressure (MAP) <70 mmHg, or SBP decrease >40 mmHg)
   * White blood cell (WBC) >12,000 u/L or <4000 u/L or immature forms >10%
   * Platelet count <100,000 u/L
   * Altered mental status with Glasgow Coma Score (GCS) <15
   * Hypoxemia (Pulse Oximetry Level <95)
   * Ileus
   * Significant edema or positive fluid balance
   * Decreased capillary refill or mottling
   * Hyperglycemia (plasma glucose >140 mg/dL) in the absence of diabetes
   * Plasma C-reactive protein >2 SD above the normal value
   * Plasma procalcitonin > 2 SD above the normal value
   * Arterial hypoxemia (PaO2 / FIO2 <300)
   * Acute oliguria (urine output <0.5 mL/kg/hr or 45 mmol/L for 2 hours)
   * Creatinine increase >0.5 mg/dL
   * INR >1.5 or a PTT >60 seconds
   * Plasma total bilirubin >4 mg/dl or 70 mmol/L
   * Hyperlactatemia (>1 mmol/L)

   4.2 For pediatric patients (>30 days old and <18 years old), all of the 3 following symptoms:
   * Fever or hypothermia (rectal temperature defined as >38.5 C or <35.0 C [or equivalent])
   * Tachycardia (heart rate >2 SD above the normal value for age). This could be absent in hypothermic subject.
   * Tachypnea (respiratory rate >2 SD above the normal value for age)

   AND at least one of the following parameters:
   * Altered mental status,(e.g., drowsiness, poor quality of cry, poor reaction to parent stimuli, and poor response to social overtures)
   * Systolic blood pressure <2 SD below the normal value for age OR narrow pulse pressure (<20 mmHg) OR poor perfusion (capillary refill >2 sec)
   * Hypoxemia (Pulse Oximetry Level <95)
   * White blood cell >15,000 u/L or <5,000 u/L or immature forms >10%.
5. Informed Consent has been obtained.

Exclusion Criteria:

* Admitted to the study site hospital for this current episode for more than 24 hours before enrollment.
* Hospitalized for this current episode for more than 72 hours at another primary/referring hospital.
* Prior to this current episode, the subject was admitted to any hospital within the last 30 days.
* An underlying pre-existing condition is thought to have led to or contributed to this sepsis episode. For example, sepsis is considered to be directly attributable to existing non-infectious conditions such as stroke, cardiovascular diseases, acute myocardial infarction, cancer, burn, injury, and trauma.
* Prior to enrollment, it is documented by the attending physician that hospital acquired infection is associated with the cause of the sepsis or severe sepsis.
* The subject has been enrolled into this study or another sepsis study before.

Min Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients, age 30 days on the day of enrollment with community-acquired sepsis or severe sepsis in Southeast Asia. Of the 2,250 enrolled patients, 1,125 will be adults and 1,125 will be children.
Sampling Method: Probability Sample
Enrollment: 2250 (Actual)
Dates: Start 2013-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The etiology of community-acquired sepsis and severe sepsis expressed in percentages of enrolled subjects. | Total length of time that subjects will be in the study is 28 to 35 days.

SECONDARY OUTCOMES:
The time from hospital admission to any systemic antibiotic administration. | 2 years
Percentage of initial systemic antimicrobial effective to treat the cause of the infection. | 2 years
Percentage of subjects receiving fluid challenge (giving bolus of fluid) if the patient has hypotension. | 2 years
Percentage of subjects receiving adequate ventilatory support (including percentage of subjects receiving supplemental oxygen, percentage of subjects receiving Positive-end Expiratory Pressure (PEEP). | 2 years
Percentage of subjects receiving low-volume lung-protective ventilation. | 2 years
Percentage of subjects receiving arterial blood gas evaluation). | 2 years
Percentage of subjects receiving renal replacement therapies (including hemodialysis and peritoneal dialysis). | 2 years
Percentage of subjects receiving imaging to determine source or deep foci of infection (including chest radiography, ultrasonogram, CT scan and MRI). | 2 years
Percentage of subjects receiving evaluation by scoring system. | 2 years
Percentage of subjects receiving stress prophylaxis. | 2 years
Percentage of patients receiving deep vein thrombosis (DVT) prophylaxis. | 2 years
Percentage of subjects receiving treatment in ICUs. | 2 years
28-day mortality rate. | 2 years
Percentage of subjects developing major organ dysfunction; for example ventilatory failure and renal failure. | 2 years
Risk factors associated with sepsis or severe sepsis | 2 years
Prevalence of antimicrobial resistance and its association with appropriate empirical therapy and outcomes. | 2 years
Sensitivities and specificities of selected RDTs in determining the causes of community-acquired sepsis and severe sepsis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Direk Limmathurotsakul, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (15):
- Indonesia (4):
  - Dr. Sardjito Hospital, Yogyakarta, DI Yogyakarta
  - Cipto Mangunkusumo Hospital, Jakarta, DKI Jaya
  - Universitas Hasanuddin, Makassar, South Sulawesi
  - Dr. Wahidin Soedirohusodo, Makassar, South Sulawesi
- Thailand (5):
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand, Bangkok, Bangkok
  - Pediatric Unit Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand, Bangkok, Bangkok
  - Queen Sirikit National Institute of Child Health, Bangkok, Bangkok
  - Sappasitthiprasong Hospital, Ubon Ratchathani, Changwat Ubon Ratchathani
  - Chiangrai Prachanukroh Hospital, Chiangrai, Chiangrai
- Vietnam (6):
  - National Hospital of Paediatric, Hanoi, Hanoi
  - National Hospital of Tropical Diseases, Hanoi, Hanoi
  - Children Hospital 1, Ho Chi Minh City, Ho Chi Minh City
  - Children Hospital 2, Ho Chi Minh City, Ho Chi Minh City
  - Hospital of Tropical Diseases, Ho Chi Minh City, Ho Chi Minh City
  - Hue Central Hospital, Huế, Hue City

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] World Health Organization (2008) The global burden of disease: 2004 update.
- [Background] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL; International Surviving Sepsis Campaign Guidelines Committee; American Association of Critical-Care Nurses; American College of Chest Physicians; American College of Emergency Physicians; Canadian Critical Care Society; European Society of Clinical Microbiology and Infectious Diseases; European Society of Intensive Care Medicine; European Respiratory Society; International Sepsis Forum; Japanese Association for Acute Medicine; Japanese Society of Intensive Care Medicine; Society of Critical Care Medicine; Society of Hospital Medicine; Surgical Infection Society; World Federation of Societies of Intensive and Critical Care Medicine. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Crit Care Med. 2008 Jan;36(1):296-327. doi: 10.1097/01.CCM.0000298158.12101.41. PMID 18158437
- [Background] Maitland K, Kiguli S, Opoka RO, Engoru C, Olupot-Olupot P, Akech SO, Nyeko R, Mtove G, Reyburn H, Lang T, Brent B, Evans JA, Tibenderana JK, Crawley J, Russell EC, Levin M, Babiker AG, Gibb DM; FEAST Trial Group. Mortality after fluid bolus in African children with severe infection. N Engl J Med. 2011 Jun 30;364(26):2483-95. doi: 10.1056/NEJMoa1101549. Epub 2011 May 26. PMID 21615299
- [Background] Cheng AC, West TE, Limmathurotsakul D, Peacock SJ. Strategies to reduce mortality from bacterial sepsis in adults in developing countries. PLoS Med. 2008 Aug 19;5(8):e175. doi: 10.1371/journal.pmed.0050175. PMID 18752342
- [Background] Suttinont C, Losuwanaluk K, Niwatayakul K, Hoontrakul S, Intaranongpai W, Silpasakorn S, Suwancharoen D, Panlar P, Saisongkorh W, Rolain JM, Raoult D, Suputtamongkol Y. Causes of acute, undifferentiated, febrile illness in rural Thailand: results of a prospective observational study. Ann Trop Med Parasitol. 2006 Jun;100(4):363-70. doi: 10.1179/136485906X112158. PMID 16762116
- [Background] Gasem MH, Wagenaar JF, Goris MG, Adi MS, Isbandrio BB, Hartskeerl RA, Rolain JM, Raoult D, van Gorp EC. Murine typhus and leptospirosis as causes of acute undifferentiated fever, Indonesia. Emerg Infect Dis. 2009 Jun;15(6):975-7. doi: 10.3201/eid1506.081405. PMID 19523308
- [Background] Phongmany S, Rolain JM, Phetsouvanh R, Blacksell SD, Soukkhaseum V, Rasachack B, Phiasakha K, Soukkhaseum S, Frichithavong K, Chu V, Keolouangkhot V, Martinez-Aussel B, Chang K, Darasavath C, Rattanavong O, Sisouphone S, Mayxay M, Vidamaly S, Parola P, Thammavong C, Heuangvongsy M, Syhavong B, Raoult D, White NJ, Newton PN. Rickettsial infections and fever, Vientiane, Laos. Emerg Infect Dis. 2006 Feb;12(2):256-62. doi: 10.3201/eid1202.050900. PMID 16494751
- [Background] Hoa NT, Diep TS, Wain J, Parry CM, Hien TT, Smith MD, Walsh AL, White NJ. Community-acquired septicaemia in southern Viet Nam: the importance of multidrug-resistant Salmonella typhi. Trans R Soc Trop Med Hyg. 1998 Sep-Oct;92(5):503-8. doi: 10.1016/s0035-9203(98)90891-4. PMID 9861362
- [Background] Wijedoru LP, Kumar V, Chanpheaktra N, Chheng K, Smits HL, Pastoor R, Nga TV, Baker S, Wuthiekanun V, Peacock SJ, Putchhat H, Parry CM. Typhoid fever among hospitalized febrile children in Siem Reap, Cambodia. J Trop Pediatr. 2012 Feb;58(1):68-70. doi: 10.1093/tropej/fmr032. Epub 2011 Apr 20. PMID 21508082
- [Background] Suputtamongkol Y, Hall AJ, Dance DA, Chaowagul W, Rajchanuvong A, Smith MD, White NJ. The epidemiology of melioidosis in Ubon Ratchatani, northeast Thailand. Int J Epidemiol. 1994 Oct;23(5):1082-90. doi: 10.1093/ije/23.5.1082. PMID 7860160
- [Background] Limmathurotsakul D, Wongratanacheewin S, Teerawattanasook N, Wongsuvan G, Chaisuksant S, Chetchotisakd P, Chaowagul W, Day NP, Peacock SJ. Increasing incidence of human melioidosis in Northeast Thailand. Am J Trop Med Hyg. 2010 Jun;82(6):1113-7. doi: 10.4269/ajtmh.2010.10-0038. PMID 20519609
- [Background] Bhengsri S, Baggett HC, Jorakate P, Kaewpan A, Prapasiri P, Naorat S, Thamthitiwat S, Tanwisaid K, Chantra S, Salika P, Dejsirilert S, Peruski LF, Maloney SA. Incidence of bacteremic melioidosis in eastern and northeastern Thailand. Am J Trop Med Hyg. 2011 Jul;85(1):117-20. doi: 10.4269/ajtmh.2011.11-0070. PMID 21734135
- [Background] Hashairi F, Hasan H, Azlan K, Deris ZZ. An eight-year review of blood culture and susceptibility among sepsis cases in an emergency department in Northeastern Malaysia. Trop Biomed. 2011 Dec;28(3):599-605. PMID 22433889
- [Background] Deen J, von Seidlein L, Andersen F, Elle N, White NJ, Lubell Y. Community-acquired bacterial bloodstream infections in developing countries in south and southeast Asia: a systematic review. Lancet Infect Dis. 2012 Jun;12(6):480-7. doi: 10.1016/S1473-3099(12)70028-2. PMID 22632186
- [Background] Angkasekwinai N, Rattanaumpawan P, Thamlikitkul V. Epidemiology of sepsis in Siriraj Hospital 2007. J Med Assoc Thai. 2009 Mar;92 Suppl 2:S68-78. PMID 19562989
- [Background] Dellinger RP, Carlet JM, Masur H, Gerlach H, Calandra T, Cohen J, Gea-Banacloche J, Keh D, Marshall JC, Parker MM, Ramsay G, Zimmerman JL, Vincent JL, Levy MM; Surviving Sepsis Campaign Management Guidelines Committee. Surviving Sepsis Campaign guidelines for management of severe sepsis and septic shock. Crit Care Med. 2004 Mar;32(3):858-73. doi: 10.1097/01.ccm.0000117317.18092.e4. PMID 15090974
- [Background] Phua J, Koh Y, Du B, Tang YQ, Divatia JV, Tan CC, Gomersall CD, Faruq MO, Shrestha BR, Gia Binh N, Arabi YM, Salahuddin N, Wahyuprajitno B, Tu ML, Wahab AY, Hameed AA, Nishimura M, Procyshyn M, Chan YH; MOSAICS Study Group. Management of severe sepsis in patients admitted to Asian intensive care units: prospective cohort study. BMJ. 2011 Jun 13;342:d3245. doi: 10.1136/bmj.d3245. PMID 21669950
- [Background] Khwannimit B, Bhurayanontachai R. The epidemiology of, and risk factors for, mortality from severe sepsis and septic shock in a tertiary-care university hospital setting. Epidemiol Infect. 2009 Sep;137(9):1333-41. doi: 10.1017/S0950268809002027. Epub 2009 Feb 4. PMID 19192320
- [Background] Kanoksil M, Jatapai A, Peacock SJ, Limmathurotsakul D. Epidemiology, microbiology and mortality associated with community-acquired bacteremia in northeast Thailand: a multicenter surveillance study. PLoS One. 2013;8(1):e54714. doi: 10.1371/journal.pone.0054714. Epub 2013 Jan 18. PMID 23349954
- [Background] Hof H. An update on the medical management of listeriosis. Expert Opin Pharmacother. 2004 Aug;5(8):1727-35. doi: 10.1517/14656566.5.8.1727. PMID 15264987
- [Background] Temple ME, Nahata MC. Treatment of listeriosis. Ann Pharmacother. 2000 May;34(5):656-61. doi: 10.1345/aph.19315. PMID 10852095
- [Background] Hof H. Listeriosis: therapeutic options. FEMS Immunol Med Microbiol. 2003 Apr 1;35(3):203-5. doi: 10.1016/S0928-8244(02)00466-2. PMID 12648838
- [Background] Personal communication with Professor Jeremy Farrar, Director, Oxford University Clinical Research Unit, Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam.
- [Background] West TE CN, Chierakul W, Limmathurotsakul D, Wuthiekanun V, Myers ND, Emond MJ, Wurfel MM, Hawn TR, Peacock SJ, Skerrett SJ. A hypofunctional TLR5 is genetic variant is associated with survival in meliodosis. 2011
- [Derived] Lie KC, Lau CY, Van Vinh Chau N, West TE, Limmathurotsakul D; for Southeast Asia Infectious Disease Clinical Research Network. Utility of SOFA score, management and outcomes of sepsis in Southeast Asia: a multinational multicenter prospective observational study. J Intensive Care. 2018 Feb 14;6:9. doi: 10.1186/s40560-018-0279-7. eCollection 2018. PMID 29468069
- [Derived] Southeast Asia Infectious Disease Clinical Research Network. Causes and outcomes of sepsis in southeast Asia: a multinational multicentre cross-sectional study. Lancet Glob Health. 2017 Feb;5(2):e157-e167. doi: 10.1016/S2214-109X(17)30007-4. PMID 28104185